CLINICAL TRIAL: NCT02970708
Title: Efficacy and Safety of Eyetronix Flicker Glasses to the Treatment of Anisometropic Amblyopia in Chinese Children
Brief Title: Efficacy and Safety of Eyetronix Flicker Glasses to the Treatment of Anisometropic Amblyopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YFZX2016001
Record Dates: First submitted 2016-11-17; First posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Amblyopia, Anisometropic
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EFG group (Experimental): amblyopia in EFG group will receive Eyetronix Flicker Glassess treatment.
  Interventions: Device: EFG group
- Patching group (Active Comparator): amblyopia in patching group will receive patching treatment.
  Interventions: Device: Patching group

INTERVENTIONS:
Device: EFG group — 88 anisometropic amblyopia will be recruited to receive Eyetronix Flicker Glasses treatment.
  Arms: EFG group
Device: Patching group — 88 anisometropic amblyopia will be recruited to receive patching treatment.
  Arms: Patching group

SUMMARY:
To evaluate the efficacy and safety of Eyetronix Flicker Glassess therapy in treating anisometropic amblyopia.

DETAILED DESCRIPTION:
A total of 176 children with anisometropic amblyopia, aged 4 to 13 years, will randomize to receive patching or Eyetronix Flicker Glasses treatment in a 1:1 ratio.Eyetronix Flicker Glasses, a lightweight spectacle frame with liquid crystal lenses that provide direct square-wave alternating occlusion, will be used at a pre-programmed temporal frequency. Patching is a traditional treatment of amblyopia. The best corrected visual acuity, contrast sensitivity, binocular function,visual evoked potential and functional MRI will be measured at baseline and follow-up visits to assess the improvement of amblyopia.Feedback information from the questionnaires will be used to evaluate the compliance and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. aged from 4 to 13 years old
2. the best corrected visual acuity in the amblyopic eye is no more than 0.1logMAR, with two lines or more of difference between the two eyes
3. anisometropia is defined as an inter-ocular spherical refractive error difference of 1.00 D or more or a cylindrical difference of 1.50 D or more.
4. no amblyopia treatment one month prior to the study except refractive correction.
5. myopia is less than -6.00D or hyperopia is less than +9.00D, strabismus was less than 20 prism diopters
6. willing to participate in this study and be able to follow up on time

Exclusion Criteria:

1. ocular disease and other disease that have an influence on the visual acuity
2. history of ocular surgery that have an influence on the visual acuity
3. the patient is receiving other amblyopia treatment except refractive correction
4. a family or personal history of seizures
5. the patient is using some medicine that may have an influence on visual acuity

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
best corrected visual acuity | 6 months
  have an improvement of best corrected visual acuity in the amblyopic eyes

SECONDARY OUTCOMES:
stereocuity | 6 months
  have an improvement of stereocuity in the amblyopic eyes
contrast sensitivity function | 6 months
  have an improvement of contrast sensitivity in the amblyopic eyes
visual evoked potential | 6 months
  P100 latency decrease and N75-P100 amplitude increase in the amblyopic eye.
functional MRI | 6 months
  the visual cortex activity have an improvement
best corrected visual acuity | a year and a half
  have an improvement of best corrected visual acuity in the amblyopic eyes

IPD SHARING:
Plan to Share IPD: Undecided